CLINICAL TRIAL: NCT02261766
Title: Detection of Atrial Fibrillation, -Evaluation of 5 Days Holter and 30 Days Thumb-ECG for Detection of Atrial Fibrillation in Stroke Patients
Brief Title: Evaluation of 5 Days Holter and 30 Days Thumb-ECG for Detection of Atrial Fibrillation in Stroke Patients
Acronym: EHOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Karsten Overgaard, Medical Doctor, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EHOT001
Record Dates: First submitted 2014-10-01; First posted 2014-10-10 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Holter monitoring and Thumb ECG — 5 days holtermonitoring and 30 days 30 seconds twice daily thumb ECG recording

SUMMARY:
This study will compare the two methods 5 days holtermonitoring and 30 days thumb electrocardiogram for detection of atrial fibrillation in stroke patients

DETAILED DESCRIPTION:
Patients with a newly stroke will be examined with both 5 day holter monitoring and 30 days thumb ECG at the same time. The detection rates of the two methods will be compared

ELIGIBILITY:
Inclusion Criteria:

* stroke or TIA within the last 3 months verified by a CT or a MR scan or unequivocal symptoms and old infarcts visualised on CT or MR
* age 65 or above
* patients able to handle the thumb-ECG
* written informed consent

Exclusion Criteria:

* earlier diagnose of atrial fibrillation
* pacemaker or ICD device
* stroke induced by trauma, infection or surgery procedure
* carotid stenosis of more than 60%

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation detection rate on Thumb-ECG | 1 month

SECONDARY OUTCOMES:
Atrial fibrillation detection rate on holtermonitoring | 5 days
Time to detection of atrial fibrillation on holter | 5 days
Time to detection af atrial fibrillation on thumb-ECG | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Derived] Poulsen MB, Binici Z, Dominguez H, Soja AM, Kruuse C, Hornnes AH, Rasmussen RS, Overgaard K. Performance of short ECG recordings twice daily to detect paroxysmal atrial fibrillation in stroke and transient ischemic attack patients. Int J Stroke. 2017 Feb;12(2):192-196. doi: 10.1177/1747493016669883. Epub 2016 Sep 30. PMID 27694312